CLINICAL TRIAL: NCT03976518
Title: Phase II, Open-label Study of Atezolizumab in a Cohort of Pretreated, Advanced Non-small Cell Lung Cancer (NSCLC) Patients With Rare Histological Subtypes (CHANCE Trial).
Brief Title: Atezolizumab in Advanced Non-small Cell Lung Cancer With Rare Histologies (CHANCE Trial)
Acronym: CHANCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Collaborators: AOU S.Orsola Malpighi-Unit of Oncologic Molecular and Transplantations Pathology (Unknown); Istituto Toscano Tumori (Other); YGHEA, CRO Division of Ecol Studio spa (Industry); Iqvia Pty Ltd (Industry); AOU S. Orsola Malpighi - Clinical Trial Office (Unknown); Silvano Chiapparoli Logistica SpA (Unknown); Roche SpA (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOIRC-02-2018
Record Dates: First submitted 2019-05-31; First posted 2019-06-06 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Advanced Non-Small Cell Lung Cancer; NSCLC Rare Histological Subtypes
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: Single-arm, open label clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATEZOLIZUMAB (Experimental): Atezolizumab will be administered at a flat dose of 1200 mg by intravenous route. Atezolizumab will be delivered in 250-mL 0.9% NaCl (sodium chloride) intravenous (IV) infusion bags. The administration will be repeated every 3 weeks (21 [± 3] days). The initial dose will be delivered over 60 (± 15) minutes. In case the first infusion is tolerated without any infusion-associated AEs the second infusion may be delivered over 30 (± 10) minutes. If the second 30 minutes infusion is well tolerated all the subsequent infusions may be administered over 30 (± 10) minutes. The treatment will be continued until disease progression, intolerable toxicity, patient refusal or Investigator's decision or any criterion for withdrawal from the trial or trial drug is fulfilled.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered on Day 1 every 21 days (+/- 3 days).

SUMMARY:
This study is aimed to explore the antitumor activity and the safety profile of atezolizumab in pretreated advanced NSCLC patients with rare histological subtypes.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced, relapsed or metastatic non-small cell lung cancer (NSCLC) - stage IIIB/IV according to 7th International Association for the Study of Lung Cancer (IASLC) classification
* Histologically confirmed diagnosis of non-small cell lung cancer (NSCLC) with rare histological subtype, according to World Health Organization (WHO) 2015 classification. Histologic subtype variants to be enrolled into the study include: colloid adenocarcinoma (or adenocarcinoma with colloid features); fetal adenocarcinoma (or adenocarcinoma with fetal features); large cell carcinoma (LCC); sarcomatoid carcinoma (pleomorphic, spindle cell, and/or giant cell carcinoma, carcinosarcoma, pulmonary blastoma); salivary gland-type tumors (mucoepidermoid carcinoma, adenoid cystic carcinoma, epithelial-myoepithelial carcinoma), other and unclassified carcinomas (lymphoepithelioma-like carcinoma, NUT-nuclear protein in testis-carcinoma)
* Availability of tumor sample (material obtained from core-biopsy or surgical specimen) for central pathology revision is mandatory
* Availability of a formalin-fixed, paraffin-embedded (FFPE) tumor block or 7-10 unstained tumor slides suitable for PD-L1 expression assessment is mandatory. The assessment of PD-L1 expression will be performed by using both SP-142 and SP-263 antibody assays. The collection of tumor sample should be performed before patients are enrolled into the study
* Male and female and ≥ 18 years of age
* Life expectancy ≥ 12 weeks
* Progressive disease after or during at least one previous standard chemotherapy line
* Measurable disease per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1); clear radiological evidence of disease progression after previous treatment has to be documented
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 2
* Patients with treated brain metastases with stable lesions for at least 2 weeks either off steroids or on a stable dose or decreasing dose of steroids (≤ 10 mg prednisone or equivalent daily) will be enrolled. Radiotherapy must have been completed a minimum of 14 days prior to registration, and patients must have recovered from adverse events (AEs) related to radiotherapy to < grade 1 (except alopecia)
* For Females: must be postmenopausal for at least 1 year before the screening visit, or are surgically sterile or not sexually active. Women of childbearing potential (WOCBP) must use 2 effective methods of contraception with a failure rate of less than 1% per year, during the entire study treatment period and for a period of 5 months after the last dose of study drug, or agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. WOCBP must have a negative serum pregnancy test during the screening period
* Adequate haematological function defined by white blood cell (WBC) count ≥2,500/mm3 with absolute neutrophil count (ANC) ≥1,500/mm3, platelet count - Adequate hepatic function defined by a total bilirubin ≤ 1.5 x the upper limit of normal (ULN) range (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL), serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN (≤ 5 if liver function test elevations are due to liver metastases)
* Adequate renal function defined by a serum creatinine ≤ 1.5 x ULN or an estimated creatinine clearance of ≥ 30 mL/minute for patients with creatinine levels above institutional limits (if using the Cockcroft-Gault formula)
* Stable medical condition, including the absence of acute exacerbations of chronic illnesses, serious infections, or major surgery within 4 weeks before registration, and otherwise noted in other inclusion/exclusion criteria
* Recovered (i.e., ≤ Grade 1 toxicity) from effects of prior anticancer therapy, except alopecia
* Ability to comply with protocol requirements
* The patient is able to provide written informed consent. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that the patient may withdraw consent at any time without prejudice to future medical care.

Exclusion Criteria:

* Prior treatment with Atezolizumab or any other immunotherapy agents (anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways)
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
* Concurrent anticancer treatment, immune therapy, or cytokine therapy, except for erythropoietin
* Major surgery for any reason within 4 weeks (or 2 weeks for minor surgery) from registration and/or if the subject has not fully recovery from the surgery within 4 weeks of registration
* Subjects receiving immunosuppressive agents such as steroids for any reason should be tapered off these drugs before initiation of the trial treatment. Corticosteroid therapy with a dose ≤ 10 mg prednisone or equivalent will be allowed. Note:

  1. Subjects receiving bisphosphonates or denosumab are eligible provided treatment was initiated at least 14 days before first dose of trial treatment
  2. Previous or ongoing administration of systemic steroids for the management of an acute allergic phenomenon is acceptable as long as it is anticipated that the administration of steroids will be completed in 14 days, or that the daily dose after 14 days will be ≤10 mg per day of equivalent prednisone
* Persisting toxicity related to prior therapy of grade >1 according to National Cancer Institute - Common Terminology Criteria Adverse Event (NCI-CTCAE) v. 4.03
* Known severe hypersensitivity reactions to chimeric or monoclonal antibodies, fusion proteins (grade ≥3 NCI-CTCAE v. 4.03)
* Patients with untreated, symptomatic and/or progressive brain metastases, or with carcinomatous meningitis. Subjects with brain metastases are eligible if metastases have been treated and there is no clinical evidence of progression for [lowest minimum is 2 weeks or more] after treatment is complete and within 28 days prior to the first dose of atezolizumab administration. In addition, subjects must be either off corticosteroids, or on a stable or decreasing dose of 10 mg daily prednisone (or equivalent)
* History of autoimmune disease, including, but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis or glomerulonephritis. Subjects with diabetes mellitus type I, hypothyroidism only requiring hormone replacement or controlled hyperthyroidism, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enrol. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of registration will be not eligible. Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10 mg or 10 mg equivalent prednisone per day. Topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption) are permitted
* Any medical condition requiring a systemic corticosteroid treatment at doses >10 mg prednisone per day or equivalent or other immunosuppressive therapies
* Other concurrent neoplasms
* Prior organ transplantation, including allogenic stem-cell transplantation
* Any medical condition, within 6 months before receiving the first dose of study drug, considered relevant by Investigator. Chronic stable atrial fibrillation on stable anticoagulant therapy is allowed. Patients who present particular clinical conditions or relevant comorbidity may be enrolled into the study upon discussion with the Study Coordinator
* Known human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)
* Any positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection
* Infection requiring intravenous (IV) antibiotic therapy or other serious infection within 14 days before the first dose of study drug
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Active tuberculosis
* Pregnancy or breastfeeding
* Vaccination within 4 weeks of the first dose of atezolizumab and while on trial is prohibited except for administration of inactivated vaccines (for example, inactivated flu vaccines)
* Unwilling or unable to comply with the protocol or cooperate fully with the investigator and site personnel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | From the start of treatment (baseline) to the progression of disease (PD) or trial discontinuation whichever occurs first, assessed up to 24 months.
  Proportion of patients presenting Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) based on the Investigator's assessment according to standard RECIST criteria v.1.1.

SECONDARY OUTCOMES:
Treatment Safety based on Adverse Events Frequency and Safety | From the treatment start to 90 days after the administration of the last treatment dose. The outcome is assessed up to a maximum of 27 months.
  Frequency and Severity of Adverse Events, the latter measured by each Investigator according to NCI Common Terminology Criteria for Adverse Events, version 4.03
Objective Response Rate (ORR) | From the start of treatment (baseline) to the progression or stability of disease assessed up to 24 months.
  Proportion of patients presenting Complete Response (CR) or Partial Response (PR) based on Investigator's assessment according to standard RECIST criteria v.1.1.
Overall Survival (OS) | From the date of enrollment to the date of death from any cause. The survival follow-up will continue until 6 months after the last subject receives the last dose of atezolizumab
  Time from enrollment until death from any cause
Time To Progression (Time To Progression) | From the date of enrollment to the date of objective tumor progression assessed up to 24 months.
  Time from enrollment until objective tumor progression assessed by the Investigators according to standard RECIST criteria v.1.1.
Progression Free Survival (PFS) | From the date of enrollment to the date of objective disease progression or death assessed up to 24 months.
  Time from enrollment until objective tumor progression or death from any cause or the last date the patient was known-to be progression free or alive

OTHER OUTCOMES:
Duration of Response (DoR) | From the time of documentation of tumor response to the time of disease progression assessed up to 24 months after baseline
  Time from documentation of tumor response (CR or PR) to tumor progression assessed by the Investigators according to standard RECIST 1.1 criteria
Time to Response | The occurrence of a response will be assessed from baseline up to 24 months
  Time from the baseline to a documented tumor response (CR or PR) assessed by the Investigators according to standard RECIST criteria v.1.1.
Tumor shrinkage in target lesions | Up to 36 months from the treatment start
  Tumor shrinkage will be determined based on the change in the sum of the longest diameter of target lesions at each time point
PD-L1 marker expression on tumor tissue | Up to 48 months from the treatment start
  Archival tumor tissue (FFPE tumor block or 7-10 unstained slides) will be assessed for determination of PD-L1 status on tumor cells by using both SP-142 and SP-263 antibody assays
Predictable value of PD-L1 tumor expression on tumor response | Up to 48 months from the treatment start
  Statistical analysis will be performed to evaluate the role of PD-L1 expression on tumor cells as predictive biomarker of tumor response
PD-L1 marker expression on Tumor Infiltrating Lymphocytes (TILs) | Up to 48 months from the treatment start
  Archival tumor tissue (FFPE tumor block or 7-10 unstained slides) will be assessed for determination of PD-L1 status on immune cells by using both SP-142 and SP-263 antibody assays
Predictable value of PD-L1 TILs expression on tumor response | Up to 48 months from the treatment start
  Statistical analysis will be performed to evaluate the role of PD-L1 expression on immune cells as predictive biomarker of tumor response
Correlation between PD-L1 expression both on tumor cells and on immune cells | Up to 48 months from the treatment start
  Correlation analysis will be performed with the aim to evaluate PD-L1 expression on both tumor cells and immune cells
Accuracy of antibody assays SP-142 and SP-263 | Up to 48 months from the treatment start
  It will be evaluated the accuracy of both antibody assays and statistical analysis will be performed to investigate their predictive value of response

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ardizzoni, MD, Principal Investigator — Dept Oncology-Haematology - S.Orsola-Malpighi Hospital - Bologna - Italy; Francesco Gelsomino, MD, Study Chair — Dept Oncology-Haematology - S.Orsola-Malpighi Hospital - Bologna - Italy
Locations (10):
- Italy (10):
  - UO Oncologia Polmonare - AOU S. Luigi Gonzaga, Orbassano, Torino
  - UO di Oncologia Medica - Azienda Ospedaliero-Universitaria S. Orsola Malpighi, Bologna
  - Dipartimento di Oncologia Medica - Azienda Ospedaliera S.Croce e Carle Cuneo - Ospedale Carle, Cuneo
  - S.S. di Oncologia Medica toraco-polmonare - Fondazione IRCCS - Istituto Nazionale Tumori, Milan
  - U.O.C Pneumologia ad Indirizzo Oncologico -AORN Ospedali dei Colli Monaldi-Cotugno-CTO, Napoli
  - UOC di Oncologia Medica 2 - IOV Istituto Oncologico Veneto, Padua
  - UOC di Oncologia Medica - Azienda Ospedaliero Universitaria di Parma, Parma
  - US di Oncologia Medica - A.O. di Perugia, Perugia
  - S.C. di Oncologia Medica - IFO - Istituto Regina Elena, Roma
  - UOC di Oncologia Medica - Azienda Sanitaria Universitaria Integrata di Udine, Udine

REFERENCES:
- [Background] Champiat S, Dercle L, Ammari S, Massard C, Hollebecque A, Postel-Vinay S, Chaput N, Eggermont A, Marabelle A, Soria JC, Ferte C. Hyperprogressive Disease Is a New Pattern of Progression in Cancer Patients Treated by Anti-PD-1/PD-L1. Clin Cancer Res. 2017 Apr 15;23(8):1920-1928. doi: 10.1158/1078-0432.CCR-16-1741. Epub 2016 Nov 8. PMID 27827313
- [Background] Ferlay J, Steliarova-Foucher E, Lortet-Tieulent J, Rosso S, Coebergh JW, Comber H, Forman D, Bray F. Cancer incidence and mortality patterns in Europe: estimates for 40 countries in 2012. Eur J Cancer. 2013 Apr;49(6):1374-403. doi: 10.1016/j.ejca.2012.12.027. Epub 2013 Feb 26. PMID 23485231
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2016. CA Cancer J Clin. 2016 Jan-Feb;66(1):7-30. doi: 10.3322/caac.21332. Epub 2016 Jan 7. PMID 26742998
- [Background] Chemotherapy in non-small cell lung cancer: a meta-analysis using updated data on individual patients from 52 randomised clinical trials. Non-small Cell Lung Cancer Collaborative Group. BMJ. 1995 Oct 7;311(7010):899-909. PMID 7580546
- [Background] Scagliotti GV, Parikh P, von Pawel J, Biesma B, Vansteenkiste J, Manegold C, Serwatowski P, Gatzemeier U, Digumarti R, Zukin M, Lee JS, Mellemgaard A, Park K, Patil S, Rolski J, Goksel T, de Marinis F, Simms L, Sugarman KP, Gandara D. Phase III study comparing cisplatin plus gemcitabine with cisplatin plus pemetrexed in chemotherapy-naive patients with advanced-stage non-small-cell lung cancer. J Clin Oncol. 2008 Jul 20;26(21):3543-51. doi: 10.1200/JCO.2007.15.0375. Epub 2008 May 27. PMID 18506025
- [Background] Sandler A, Gray R, Perry MC, Brahmer J, Schiller JH, Dowlati A, Lilenbaum R, Johnson DH. Paclitaxel-carboplatin alone or with bevacizumab for non-small-cell lung cancer. N Engl J Med. 2006 Dec 14;355(24):2542-50. doi: 10.1056/NEJMoa061884. PMID 17167137
- [Background] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leiby MA, Lubiniecki GM, Shentu Y, Rangwala R, Brahmer JR; KEYNOTE-024 Investigators. Pembrolizumab versus Chemotherapy for PD-L1-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2016 Nov 10;375(19):1823-1833. doi: 10.1056/NEJMoa1606774. Epub 2016 Oct 8. PMID 27718847
- [Background] Azzoli CG, Baker S Jr, Temin S, Pao W, Aliff T, Brahmer J, Johnson DH, Laskin JL, Masters G, Milton D, Nordquist L, Pfister DG, Piantadosi S, Schiller JH, Smith R, Smith TJ, Strawn JR, Trent D, Giaccone G; American Society of Clinical Oncology. American Society of Clinical Oncology Clinical Practice Guideline update on chemotherapy for stage IV non-small-cell lung cancer. J Clin Oncol. 2009 Dec 20;27(36):6251-66. doi: 10.1200/JCO.2009.23.5622. Epub 2009 Nov 16. PMID 19917871
- [Background] Peters S, Adjei AA, Gridelli C, Reck M, Kerr K, Felip E; ESMO Guidelines Working Group. Metastatic non-small-cell lung cancer (NSCLC): ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2012 Oct;23 Suppl 7:vii56-64. doi: 10.1093/annonc/mds226. No abstract available. PMID 22997455
- [Background] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Background] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Background] Herbst RS, Baas P, Kim DW, Felip E, Perez-Gracia JL, Han JY, Molina J, Kim JH, Arvis CD, Ahn MJ, Majem M, Fidler MJ, de Castro G Jr, Garrido M, Lubiniecki GM, Shentu Y, Im E, Dolled-Filhart M, Garon EB. Pembrolizumab versus docetaxel for previously treated, PD-L1-positive, advanced non-small-cell lung cancer (KEYNOTE-010): a randomised controlled trial. Lancet. 2016 Apr 9;387(10027):1540-1550. doi: 10.1016/S0140-6736(15)01281-7. Epub 2015 Dec 19. PMID 26712084
- [Background] Rittmeyer A, Barlesi F, Waterkamp D, Park K, Ciardiello F, von Pawel J, Gadgeel SM, Hida T, Kowalski DM, Dols MC, Cortinovis DL, Leach J, Polikoff J, Barrios C, Kabbinavar F, Frontera OA, De Marinis F, Turna H, Lee JS, Ballinger M, Kowanetz M, He P, Chen DS, Sandler A, Gandara DR; OAK Study Group. Atezolizumab versus docetaxel in patients with previously treated non-small-cell lung cancer (OAK): a phase 3, open-label, multicentre randomised controlled trial. Lancet. 2017 Jan 21;389(10066):255-265. doi: 10.1016/S0140-6736(16)32517-X. Epub 2016 Dec 13. PMID 27979383
- [Background] Peters S, Gettinger S, Johnson ML, Janne PA, Garassino MC, Christoph D, Toh CK, Rizvi NA, Chaft JE, Carcereny Costa E, Patel JD, Chow LQM, Koczywas M, Ho C, Fruh M, van den Heuvel M, Rothenstein J, Reck M, Paz-Ares L, Shepherd FA, Kurata T, Li Z, Qiu J, Kowanetz M, Mocci S, Shankar G, Sandler A, Felip E. Phase II Trial of Atezolizumab As First-Line or Subsequent Therapy for Patients With Programmed Death-Ligand 1-Selected Advanced Non-Small-Cell Lung Cancer (BIRCH). J Clin Oncol. 2017 Aug 20;35(24):2781-2789. doi: 10.1200/JCO.2016.71.9476. Epub 2017 Jun 13. PMID 28609226
- [Background] Fehrenbacher L, Spira A, Ballinger M, Kowanetz M, Vansteenkiste J, Mazieres J, Park K, Smith D, Artal-Cortes A, Lewanski C, Braiteh F, Waterkamp D, He P, Zou W, Chen DS, Yi J, Sandler A, Rittmeyer A; POPLAR Study Group. Atezolizumab versus docetaxel for patients with previously treated non-small-cell lung cancer (POPLAR): a multicentre, open-label, phase 2 randomised controlled trial. Lancet. 2016 Apr 30;387(10030):1837-46. doi: 10.1016/S0140-6736(16)00587-0. Epub 2016 Mar 10. PMID 26970723
- [Background] Zhang J, Sun J, Liang XL, Lu JL, Luo YF, Liang ZY. Differences between low and high grade fetal adenocarcinoma of the lung: a clinicopathological and molecular study. J Thorac Dis. 2017 Jul;9(7):2071-2078. doi: 10.21037/jtd.2017.07.14. PMID 28840008
- [Background] de Kock L, Bah I, Wu Y, Xie M, Priest JR, Foulkes WD. Germline and Somatic DICER1 Mutations in a Well-Differentiated Fetal Adenocarcinoma of the Lung. J Thorac Oncol. 2016 Mar;11(3):e31-3. doi: 10.1016/j.jtho.2015.09.012. Epub 2015 Dec 10. PMID 26886166
- [Background] Rossi G, Mengoli MC, Cavazza A, Nicoli D, Barbareschi M, Cantaloni C, Papotti M, Tironi A, Graziano P, Paci M, Stefani A, Migaldi M, Sartori G, Pelosi G. Large cell carcinoma of the lung: clinically oriented classification integrating immunohistochemistry and molecular biology. Virchows Arch. 2014 Jan;464(1):61-8. doi: 10.1007/s00428-013-1501-6. Epub 2013 Nov 13. PMID 24221342
- [Background] Pelosi G, Sonzogni A, De Pas T, Galetta D, Veronesi G, Spaggiari L, Manzotti M, Fumagalli C, Bresaola E, Nappi O, Viale G, Rosai J. Review article: pulmonary sarcomatoid carcinomas: a practical overview. Int J Surg Pathol. 2010 Apr;18(2):103-20. doi: 10.1177/1066896908330049. Epub 2009 Jan 4. PMID 19124452
- [Background] Roden AC, Greipp PT, Knutson DL, Kloft-Nelson SM, Jenkins SM, Marks RS, Aubry MC, Garcia JJ. Histopathologic and Cytogenetic Features of Pulmonary Adenoid Cystic Carcinoma. J Thorac Oncol. 2015 Nov;10(11):1570-5. doi: 10.1097/JTO.0000000000000656. PMID 26309189
- [Background] Salem A, Bell D, Sepesi B, Papadimitrakopoulou V, El-Naggar A, Moran CA, Kalhor N. Clinicopathologic and genetic features of primary bronchopulmonary mucoepidermoid carcinoma: the MD Anderson Cancer Center experience and comprehensive review of the literature. Virchows Arch. 2017 Jun;470(6):619-626. doi: 10.1007/s00428-017-2104-4. Epub 2017 Mar 25. PMID 28343305
- [Background] Masuya D, Haba R, Huang CL, Yokomise H. Myoepithelial carcinoma of the lung. Eur J Cardiothorac Surg. 2005 Nov;28(5):775-7. doi: 10.1016/j.ejcts.2005.08.003. Epub 2005 Sep 26. PMID 16188445
- [Background] He J, Shen J, Pan H, Huang J, Liang W, He J. Pulmonary lymphoepithelioma-like carcinoma: a Surveillance, Epidemiology, and End Results database analysis. J Thorac Dis. 2015 Dec;7(12):2330-8. doi: 10.3978/j.issn.2072-1439.2015.12.62. PMID 26793355
- [Background] Bauer DE, Mitchell CM, Strait KM, Lathan CS, Stelow EB, Luer SC, Muhammed S, Evans AG, Sholl LM, Rosai J, Giraldi E, Oakley RP, Rodriguez-Galindo C, London WB, Sallan SE, Bradner JE, French CA. Clinicopathologic features and long-term outcomes of NUT midline carcinoma. Clin Cancer Res. 2012 Oct 15;18(20):5773-9. doi: 10.1158/1078-0432.CCR-12-1153. Epub 2012 Aug 15. PMID 22896655
- [Background] Kim C, Rajan A, DeBrito PA, Giaccone G. Metastatic lymphoepithelioma-like carcinoma of the lung treated with nivolumab: a case report and focused review of literature. Transl Lung Cancer Res. 2016 Dec;5(6):720-726. doi: 10.21037/tlcr.2016.11.06. PMID 28149767
- [Background] Gounant V, Brosseau S, Naltet C, Opsomer MA, Antoine M, Danel C, Khalil A, Cadranel J, Zalcman G. Nivolumab-induced organizing pneumonitis in a patient with lung sarcomatoid carcinoma. Lung Cancer. 2016 Sep;99:162-5. doi: 10.1016/j.lungcan.2016.07.010. Epub 2016 Jul 15. PMID 27565934
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbe C, Maio M, Binder M, Bohnsack O, Nichol G, Humphrey R, Hodi FS. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res. 2009 Dec 1;15(23):7412-20. doi: 10.1158/1078-0432.CCR-09-1624. Epub 2009 Nov 24. PMID 19934295
- [Background] Nishino M, Giobbie-Hurder A, Gargano M, Suda M, Ramaiya NH, Hodi FS. Developing a common language for tumor response to immunotherapy: immune-related response criteria using unidimensional measurements. Clin Cancer Res. 2013 Jul 15;19(14):3936-43. doi: 10.1158/1078-0432.CCR-13-0895. Epub 2013 Jun 6. PMID 23743568